CLINICAL TRIAL: NCT01016587
Title: Symptom Clusters and Immune Markers in Patients With COPD
Brief Title: Symptom Clusters and Immune Markers in Patients With Chronic Obstructive Pulmonary Disease (COPD) - a Longitudinal Study
Acronym: SGIS
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Tone Rustøen, Senior Researcher, Oslo University Hospital
Other Study IDs: 2009055
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: symptoms; dyspnea; pain; fatigue; anxiety; depression; sleeplessness; genetic markers; immune markers; COPD; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Pain; Fatigue; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One foci is to perform a genome wide association study in patient with COPD to identify novel genetic markers for the patient subgroups who report different experiences with the symptom cluster of pain, fatigue, breathlessness, sleep disturbance, and depression. It is likely that genetic and immunologic factors may be involved in symptom severity and morbidity. Specifically, low levels of circulating immunoglobulins have been observed in a subset of COPD patients. Although hypogammaglobulinemia (HGG) is known to lead to frequent airway infections in other patients groups, the relationship between HGG and clinical symptoms in COPD has not been studied. The resulting knowledge can help clinicians to better identify COPD patients at particular risk for severe single and multiple symptoms.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COPD patients: Not hospitalized COPD patients, degree 2-4.

SUMMARY:
COPD patients often have a wide range of physical (e.g., dyspnea, fatigue, pain) and psychological (e.g., depression, anxiety) symptoms and various other debilitating conditions that cause considerable suffering for the individual. Unfortunately, many of the symptoms and health problems in patients with COPD are unrecognized and untreated. Due to the irreversible nature of COPD, the aim is not to cure the disease, but to reduce symptoms and improve quality of life.

Therefore, the purpose of this project is to investigate the existence and nature of symptom clusters over time in patients with COPD and their effects on patient outcomes. Since this study aims to identify possible new subgroups of patients with COPD defined by the clustering of certain symptoms, the study also aims to investigate the relationship between the clinical presentation and certain immunologic and genetic factors.

DETAILED DESCRIPTION:
The specific aims of this translational, interdisciplinary, multi-center, international research study will follow 308 COPD patients with repeated measures over 12 months, are to:

1. Explore COPD patients' symptoms, symptom clusters, and changes in symptoms and symptom clusters over time; as well as the genetic markers for subgroups of patients with different symptom clusters.
2. Identify the occurrence of HGG and assess immune function in COPD patients.
3. Explore relationships between HGG and immune function, genetic markers, symptoms, symptom clusters, health and respiratory status, frequency of exacerbations and health-related QOL.

ELIGIBILITY:
Inclusion Criteria:

* degree 2-4
* above 18 years of age
* able to read/ write/ speak Norwegian

Exclusion Criteria:

* patients who are receiving treatment for cancer
* acute exacerbations of COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 308 COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2009-11; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
symptom clusters in patients with COPD | 5 times during 12 months

SECONDARY OUTCOMES:
Evaluate potential candidate genes in relation to symptom clusters and investigate the relationship between hypogammaglobulinemia and symptoms in COPD. | 2 times during 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway